CLINICAL TRIAL: NCT01312025
Title: Randomized Controlled Trial Comparing Between The Conventional Technique of Laparoscopic Cholecystectomy and A Proposed Modified Technique
Brief Title: Conventional Versus Modified Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Other Study IDs: TIE123AR
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2009-08

CONDITIONS: Laparoscopic Cholecystectomy

ARMS (2):
- conventional laparoscopic cholecystectomy (Placebo Comparator)
  Interventions: Procedure: conventional laparoscopic cholecystectomy
- modified laparoscopic cholecystectomy (Active Comparator)
  Interventions: Procedure: modified laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: conventional laparoscopic cholecystectomy
  Arms: conventional laparoscopic cholecystectomy
Procedure: modified laparoscopic cholecystectomy
  Arms: modified laparoscopic cholecystectomy

SUMMARY:
In conventional laparoscopic cholecystectomy, the cystic duct and artery are clipped by metal clips. we propose a new method in which the cystic duct is ligated and the cystic artery is cauterized. the investigators compare both methods.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy for symptomatic gallstones

Exclusion Criteria:

* Conversion to laparotomy

Ages: 10 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult